CLINICAL TRIAL: NCT05021445
Title: Effects of Pilates Exercises on Dynamic Balance in Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/20/0212
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Elderly Population
Keywords: Elderly population, Dynamic Balance, Pilates Exercises,

STUDY DESIGN:
Intervention Model Description: each participant will be requested to draw either number one or number two from a box. number one will be allocated to group A . and number two will be allocated o group B. The group A consists of 12 elderly participants who received intervention protocol of Pilates- based exercises program in which total 12-sessions were given for thrice a week for four weeks for 50-minutes.
  Group B The group B consists of 12 elderly participants who received intervention protocol of Conventional balance training exercises in which total 12-sessions were given for thrice a week for four weeks for 50-minutes.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plates based exercise (Experimental): This will consists of 12 elderly participants who receive intervention protocol of Plates- based exercises program in which total 12-sessions will be given for thrice a week for four weeks for 50-minutes.
  Interventions: Combination Product: plates based exercises
- conventional treatment (Active Comparator): this will consists of 12 elderly participants who will receive intervention protocol of Conventional balance training exercises in which total 12-sessions will be given for thrice a week for four weeks for 50-minutes.
  Interventions: Combination Product: conventional exercises

INTERVENTIONS:
Combination Product: plates based exercises — 12 elderly participants receive intervention protocol of Plates- based exercises program total 12-sessions will be given for thrice a week for four weeks for 50-minutes.
  Arms: plates based exercise
Combination Product: conventional exercises — 12 elderly participants,intervention protocol of Conventional balance training exercises,total 12-sessions will be given for thrice a week for four weeks for 50-minutes.
  Arms: conventional treatment

SUMMARY:
To find out the effects of Plates exercises on dynamic balance in elderly population

DETAILED DESCRIPTION:
The process of age-related changes involves some kind of degenerative, gradual changes which are irreversible such as degradation of activity of cells and loss of physical adaptability. According to age-related changes such as changes in balance are specifically begins near the age 45 years-old, physical characteristics such as (flexibility, strength, balance and coordination) and sensory systems are affected which ultimately increase the chances of falls in elderly individuals. Balance can be defined as the ability of a person to control their position within the limits of base of support. Pilates is an individualized-based and low-intermediate intensity exercise that can be easily performed by the elderly . Conventional balance exercises which have rehabilitative effect in reducing risk of falls and enhancing functional ability in elderly population. Conventional balance training comprises of four components which are flexibility exercises, strength training, postural control exercise and endurance training.The objective of the study IS to find out the effects of Pilates exercises on dynamic balance in elderly population. The Twenty-four participants will be recruited and divided into two equal groups randomly. The group A(n=12) will perform Pilates-based exercises protocol for 50- minutes with 10-minutes warm-up phase, 30-minutes training phase and 10-minutes for cool-down phase, thrice a week for four week and the group B(n=12) will receive Conventional balance training exercises for 50-minutes, thrice a week for four weeks. Outcome measures will be were TUG and SPPB before and after the trial and the outcomes will be compared before and end of four weeks treatment protocol. Data will be analyze by SPSS version 21. Independent sample t- test and paired sample t-test will be utilize to compare and evaluate the effects of both approaches.

ELIGIBILITY:
Inclusion Criteria:

* Those who had history of fall in past one year.
* Elderly population who scores 45 on Berg Balance Scale.

Exclusion Criteria:

* Those elderly individuals who are suffering from any kind of disease that can affect their performance for example Osteoarthritis grade III & IV, scoliosis.
* Those elderly individuals who are suffering from any kind of visual, auditory and neural or vestibular system disorders.
* Those elderly individuals who are unable to understand the treatment protocol.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
time up and go test | 50 minutes
  Time Up and Go is a very simple, quick, valid, reliable and an objective test which is widely clinical performance based measure used to assess and quantify the basic mobility skills. It assesses that how a person could perform series of sequential tasks during walk and turn. TUG is commonly used for the assessment of balance and it is considered to be appropriate for elderly population which is at risk of fall.

SECONDARY OUTCOMES:
Short Physical Performance Battery test | 50 minutes
  Short Physical Performance Battery test is a well defined and most commonly tool or instrument which measures the lower extremity physical performance status in elderly population. this is an objective tool which evaluates the functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Zeest hashmi, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunsky A. The Effect of Balance and Coordination Exercises on Quality of Life in Older Adults: A Mini-Review. Front Aging Neurosci. 2019 Nov 15;11:318. doi: 10.3389/fnagi.2019.00318. eCollection 2019. PMID 31803048
- [Background] Deger TB, Sarac ZF, Savas ES, Akcicek SF. The Relationship of Balance Disorders with Falling, the Effect of Health Problems, and Social Life on Postural Balance in the Elderly Living in a District in Turkey. Geriatrics (Basel). 2019 May 17;4(2):37. doi: 10.3390/geriatrics4020037. PMID 31108836
- [Result] Molhemi F, Monjezi S, Mehravar M, Shaterzadeh-Yazdi MJ, Salehi R, Hesam S, Mohammadianinejad E. Effects of Virtual Reality vs Conventional Balance Training on Balance and Falls in People With Multiple Sclerosis: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Feb;102(2):290-299. doi: 10.1016/j.apmr.2020.09.395. Epub 2020 Nov 5. PMID 33161005